CLINICAL TRIAL: NCT00249340
Title: Comparison of a Brief Behavioral Weight Loss Intervention With the Weight Watchers Program
Brief Title: Brief Behavioral Weight Loss Treatment vs. Weight Watchers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2076-05
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2005-08

CONDITIONS: Obesity; Overweight
Keywords: behavioral weight loss treatment; brief behavioral treatment; commercial weight loss programs; Weight Watchers
MeSH Terms: conditions — Obesity; Overweight

INTERVENTIONS:
Behavioral: Weight Watchers
Behavioral: brief behavioral weight loss treatment
Behavioral: brief behavioral + Weight Watchers combined treatment

SUMMARY:
The purpose of this study is to compare the effectiveness of Weight Watchers, brief behavioral treatment, and a combination treatment. We hypothesize that a combination treatment will achieve greater weight losses than Weight Watchers alone.

DETAILED DESCRIPTION:
Weight Watchers is a popular nonmedical commercial weight loss program. Recent studies suggest that people enrolled in Weight Watchers lose approximately 3-5 kg in 6 months of treatment. These outcomes are substantially lower than average weight losses achieved in 6 months if university/hospital-based standard behavioral treatment (approximately 10 kg). However, standard behavioral weight loss programs are expensive and have limited accessibility to most people seeking weight loss. Therefore, the purpose of the current study is to investigate whether enhancing Weight Watchers by adding an 8-week group-based behavioral weight loss program prior to participation in Weight Watchers will improve weight loss outcomes at 6 months.

Comparison: 6 months of Weight Watchers vs. combination treatment (2 months of standard behavioral weight loss treatment followed by 4 months of Weight Watchers) vs. 2 months of standard behavioral treatment.

ELIGIBILITY:
Inclusion Criteria:

Age 21-65 years BMI 27-45 kg/m2 Able to sign informed consent

Exclusion Criteria:

Women who are pregnant, nursing, less than 6 months postpartum, or plan to become pregnant during course of study Individuals who report a medical condition that would affect the safety and/or efficacy of a weight management program involving dietary change and physical activity (e.g., heart disease, cancer) Individuals with major psychiatric illness that would interfere with protocol adherence Individuals who are currently participating in a weight loss program or taking weight loss medication or lost >=5% of body weight during 6 months prior to screening Recent (within the past 12 months) participation in Weight Watchers

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-11; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Weight Loss

CONTACTS AND LOCATIONS:
Overall Officials: Rena R Wing, PhD, Principal Investigator — The Miriam Hospital; Angela M Pinto, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control and Diabetes Research Center/The Miriam Hospital, Providence, Rhode Island, United States